CLINICAL TRIAL: NCT02855164
Title: A Randomized, Double-blind, Placebo Controlled, 3- Part, Adaptive Design, Multicenter Study to Assess Safety, Tolerability and Efficacy of Tropifexor (LJN452) in Patients With Non-alcoholic Steatohepatitis (NASH): FLIGHT-FXR
Brief Title: Study of Safety and Efficacy of Tropifexor (LJN452) in Patients With Non-alcoholic Steatohepatitis (NASH)
Acronym: FLIGHT-FXR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLJN452A2202; 2015-005215-33 (EudraCT Number)
Record Dates: First submitted 2016-07-20; First posted 2016-08-04 (Estimated); Results first posted 2021-07-29 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Non-alcoholic Steatohepatitis (NASH)
Keywords: LJN452; non-alcoholic steatohepatitis; NASH; phase 2; adaptive design; randomized
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — tropifexor

STUDY DESIGN:
Intervention Model Description: This was a randomized, double-blind, placebo-controlled, multicenter, parallel-group, dose finding, 3-part (Parts A, B, and C), adaptive design study to assess the safety, tolerability, and efficacy of six doses of tropifexor as compared to placebo in subjects with NASH. Each study part had a screening period followed by a double-blind, randomized, treatment period, and a post-treatment follow-up period.
  This study was extended based on safety and efficacy results in Part A and available long-term toxicology coverage; Part C was added to explore 48 weeks of treatment at higher doses with paired biopsies in F2/3 NASH patients.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- LJN452 10 μg (Experimental): Tropifexor (LJN452) Part A
  Interventions: Drug: Tropifexor (LJN452)
- LJN452 30 μg (Experimental): Tropifexor (LJN452) Part A
  Interventions: Drug: Tropifexor (LJN452)
- LJN452 60 μg (Experimental): Tropifezor (LJN452) Parts A + B
  Interventions: Drug: Tropifexor (LJN452)
- LJN452 90 μg (Experimental): Tropifexor (LJN452) Parts A + B
  Interventions: Drug: Tropifexor (LJN452)
- Placebo A+ B (Placebo Comparator): Placebo Parts A + B
  Interventions: Drug: Placebo
- LJN452 140 μg (Experimental): Tropifexor (LJN452) Part C
  Interventions: Drug: Tropifexor (LJN452)
- LJN452 200 μg (Experimental): Tropifexor (LJN452) Part B
  Interventions: Drug: Tropifexor (LJN452)
- Placebo C (Placebo Comparator): Placebo Part C
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tropifexor (LJN452) — Comparison of different doses of drug
  Arms: LJN452 10 μg; LJN452 140 μg; LJN452 200 μg; LJN452 30 μg; LJN452 60 μg; LJN452 90 μg
Drug: Placebo — Comparator
  Arms: Placebo A+ B; Placebo C

SUMMARY:
The purpose of the study was to assess the effects of different doses of tropifexor (LJN452) with respect to safety, tolerability, and on markers of liver inflammation in patients with NASH

DETAILED DESCRIPTION:
Part A In Part A, 77 subjects were randomized at baseline to receive tropifexor (10 μg, 30 μg, 60 μg or 90 μg) or placebo (Arms A, B, C, D and E) for 12 weeks. After ≥ 90% of the subjects from Part A completed 8 weeks of treatment, the first interim analysis of all Part A data was performed and the Data Monitoring Committee (DMC) recommended evaluation of 90 μg tropifexor (safe andefficacious) in Part B. The treatment arms of Part A were completed through Week 16 without adaptation.

Part B Randomization for Part B was started after the DMC recommendations on the dose to be used in Part B were implemented by the sponsor. As planned in the study protocol, since the first interim analysis selected one active dose (90 μg) to be tested in Part B, one of the other originally planned active treatment arms (60 μg) was included with a smaller sample size to confirm the earlier findings of this dose observed in Part A. Therefore, in Part B, 121 subjects, were randomized at baseline to receive tropifexor (90 μg and 60 μg) or placebo (Arms F, G and H) for 12 weeks.

Part C was introduced as a result of the DMC recommendation to pursue doses > 90 μg. Randomization in Part C started once the Part B randomization was completed. In Part C, 152 subjects were randomized at baseline to receive 140 μg or 200 μg tropifexor or placebo (Arms I, J and K) for 48 weeks.

One patient was treated at 2 sites but is still only one patient. 350 total enrollment, and not 351.

ELIGIBILITY:
Inclusion Criteria:

* male/female patients, 18 years or older
* written informed consent
* Part A and B patients : presence of NASH by histological evidence (liver biopsy obtained 2 years or less prior to randomization) with fibrosis level of F1, F2 or F3 (fibrosis in the absence of cirrhosis) and no diagnosis of chronic liver disease and elevated alanine aminotransferase (ALT) OR phenotypic diagnosis based on elevated ALT, BMI and diagnosis of Type 2 diabetes mellitus (DM)
* Part C patients: presence of NASH by histological evidence (liver biopsy obtained during the Screening period or 6 months or less prior to randomization) with fibrosis level of F2 or F3 and no diagnosis of chronic liver disease

And ( All Parts):

* ALT ≥ 43 IU/L (males) or ≥ 28 IU/L (females)
* Liver fat equal to or higher than 10% by MRI

Exclusion Criteria:

* previous exposure to OCA
* patients taking prohibited medications
* patients taking the following medicines UNLESS on a stable dose (within 25% of baseline dose) for at least 1 month before randomization: (for Part C patients, dose must be stable for at least 1 month prior to biopsy through Screening : anti- diabetic medications, insulin, beta-blockers, thiazide diuretics, fibrates, statins, niacin, ezetimibe, vitamin E (if doses > 200 IU/day; doses > 800 IU/day are prohibited), thyroid hormone, psychotropic medications, estrogen or estrogen containing birth control
* pregnant or nursing (lactating) women
* current or history of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening
* uncontrolled diabetes mellitus
* new use of GLP-1 agonists such as liraglutide, exenatide, lixisenatide, albiglutide or dulaglutide within 3 months of screening
* presence of cirrhosis
* hepatic decompensation or severe liver impairment
* previous diagnosis of other forms of chronic liver disease
* patients with contraindications to MRI imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (76):
- United States (31):
  - Novartis Investigative Site, Madison, Alabama
  - Novartis Investigative Site, North Little Rock, Arkansas
  - Novartis Investigative Site, Coronado, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, Rialto, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Lonetree, Colorado
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Lakewood Rch, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Athens, Georgia
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Catonsville, Maryland
  - Novartis Investigative Site, Worcester, Massachusetts
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Jefferson City, Missouri
  - Novartis Investigative Site, Berlin, New Jersey
  - Novartis Investigative Site, Morehead City, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Hermitage, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Norfolk, Virginia
  - Novartis Investigative Site, Richmond, Virginia
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Australia (2):
  - Novartis Investigative Site, Kingswood, New South Wales
  - Novartis Investigative Site, Fitzroy, Victoria
- Austria (2):
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Canada (3):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Chicoutimi, Quebec
- France (2):
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
- Germany (5):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, New Delhi, National Capital Territory of Delhi, India
- Italy (3):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Roma
- Japan (4):
  - Novartis Investigative Site, Hatsukaichi, Hiroshima
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Saga, Saga-ken
  - Novartis Investigative Site, Izumo, Shimane
- Novartis Investigative Site, Utrecht, Netherlands
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (3):
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Nitra
- South Korea (4):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Dongjak Gu, Seoul
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Seoul
- Spain (3):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Taiwan (5):
  - Novartis Investigative Site, Kaoshiung, Taiwan
  - Novartis Investigative Site, Keelung
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Sanyal AJ, Lopez P, Lawitz EJ, Lucas KJ, Loeffler J, Kim W, Goh GBB, Huang JF, Serra C, Andreone P, Chen YC, Hsia SH, Ratziu V, Aizenberg D, Tobita H, Sheikh AM, Vierling JM, Kim YJ, Hyogo H, Tai D, Goodman Z, Schaefer F, Carbarns IRI, Lamle S, Martic M, Naoumov NV, Brass CA. Tropifexor for nonalcoholic steatohepatitis: an adaptive, randomized, placebo-controlled phase 2a/b trial. Nat Med. 2023 Feb;29(2):392-400. doi: 10.1038/s41591-022-02200-8. Epub 2023 Feb 16. PMID 36797481
- [Derived] Naoumov NV, Brees D, Loeffler J, Chng E, Ren Y, Lopez P, Tai D, Lamle S, Sanyal AJ. Digital pathology with artificial intelligence analyses provides greater insights into treatment-induced fibrosis regression in NASH. J Hepatol. 2022 Nov;77(5):1399-1409. doi: 10.1016/j.jhep.2022.06.018. Epub 2022 Jun 30. PMID 35779659
- See also: A Randomized, Patient and Investigator Blinded, Placebo Controlled, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of LMB763 in Patients With Non-alcoholic Steatohepatitis (NASH) — https://clinicaltrials.gov/ct2/show/NCT02913105?term=NASH+novartis&rank=2

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 411 subjects were screened in Parts A and B of the study together. Of these, 198 subjects were deemed eligible to participate in the study and were subsequently randomized
Pre-assignment Details: In Part A, 77 were randomized at baseline to receive tropifexor 10 μg (n=14), 30μg (n=16), 60 μg (n=16) or 90 μg (n=15) or placebo (n=16)
  In Part B, 121 were randomized at baseline to receive tropifexor 90 μg (n=70) and 60 μg (n=21) or placebo (n=30)
  780 were screened in Part C. Of these 152 met eligibility criteria and were randomized to receive tropifexor 140 μg (n=50) or 200 μg (n=51) or placebo (n=51)
Groups:
- LJN452 10 μg: 10 micrograms of Tropifexor (Part A)
- LJN452 30 μg: 30 micrograms of Tropifexor (Part A)
- LJN452 60 μg: 60 micrograms of Tropifexor (Parts A+B)
- LJN452 90 μg: 90 micrograms of Tropifexor (Parts A + B)
- Placebo A+B: Placebo A+B
- LJN452 140 μg: 140 micrograms of Tropifexor (Part C)
- LJN452 200 μg: 200 micrograms of Tropifexor (Part C)
- Placebo C: Placebo (Part C)
Period: Parts A + B (Randomized Set)
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo A+B | LJN452 140 μg | LJN452 200 μg | Placebo C
Started | 14 | 16 | 37 | 85 | 46 | 0 | 0 | 0
Completed | 14 | 16 | 36 | 77 | 45 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 8 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Period: Part C (Randomized Set)
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo A+B | LJN452 140 μg | LJN452 200 μg | Placebo C
Started | 0 | 0 | 0 | 0 | 0 | 50 | 51 | 51
Completed | 0 | 0 | 0 | 0 | 0 | 38 | 37 | 44
Not Completed | 0 | 0 | 0 | 0 | 0 | 12 | 14 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 5 | 9 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) was all subjects to whom study treatment had been assigned. Following the intent-to-treat (ITT) principle, subjects were analyzed according to the treatment they have been assigned to at randomization.
Groups:
- Placebo A+B: Placebo (Parts A+B)
- Total: Total of all reporting groups
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo A+B | LJN452 140 μg | LJN452 200 μg | Placebo C | Total
Number analyzed (Participants) | 14 | 16 | 37 | 85 | 46 | 50 | 51 | 51 | 350
Age, Categorical [Count of Participants; unit: Participants] — Population: FAS
  Participants
    Parts A + B: number analyzed (Participants) | 14 | 16 | 37 | 85 | 46 | 0 | 0 | 0 | 198
    Parts A + B: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Parts A + B: Between 18 and 65 years | 14 | 14 | 33 | 72 | 41 | 0 | 0 | 0 | 174
    Parts A + B: >=65 years | 0 | 2 | 4 | 13 | 5 | 0 | 0 | 0 | 24
    Part C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 50 | 51 | 51 | 152
    Part C: <=18 years |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
    Part C: Between 18 and 65 years |  |  |  | 0 |  | 40 | 41 | 43 | 124
    Part C: >=65 years |  |  |  | 0 |  | 10 | 10 | 8 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Full Analysis Set
  years
    Parts A + B: number analyzed (Participants) | 14 | 16 | 37 | 85 | 46 | 0 | 0 | 0 | 198
    Parts A + B | 48 (11.7) | 49 (14.4) | 50 (12.5) | 51 (13.4) | 51 (12.3) |  |  |  | 51 (12.8)
    Part C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 50 | 51 | 51 | 152
    Part C |  |  |  |  |  | 56 (11.41) | 55 (10.8) | 54 (11.0) | 55 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of participant by treatment Population: FAS
  Participants
    Parts A + B: number analyzed (Participants) | 14 | 16 | 37 | 85 | 46 | 0 | 0 | 0 | 198
    Parts A + B: Female | 9 | 7 | 20 | 47 | 21 | 0 | 0 | 0 | 104
    Parts A + B: Male | 5 | 9 | 17 | 38 | 25 | 0 | 0 | 0 | 94
    Part C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 50 | 51 | 51 | 152
    Part C: Female | 0 | 0 | 0 | 0 | 0 | 36 | 29 | 32 | 97
    Part C: Male | 0 | 0 | 0 | 0 | 0 | 14 | 22 | 19 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: FAS
  Participants
    Caucasian (Parts A + B): number analyzed (Participants) | 14 | 16 | 37 | 85 | 46 | 0 | 0 | 0 | 198
    Caucasian (Parts A + B) | 12 | 11 | 24 | 50 | 25 |  |  |  | 122
    Black (Parts A + B): number analyzed (Participants) | 14 | 16 | 37 | 85 | 46 | 0 | 0 | 0 | 198
    Black (Parts A + B) | 0 | 0 | 0 | 1 | 0 |  |  |  | 1
    Asian (Parts A + B): number analyzed (Participants) | 14 | 16 | 37 | 85 | 46 | 0 | 0 | 0 | 198
    Asian (Parts A + B) | 2 | 5 | 12 | 31 | 20 |  |  |  | 70
    Pacific Islander (Parts A + B): number analyzed (Participants) | 14 | 16 | 37 | 85 | 46 | 0 | 0 | 0 | 198
    Pacific Islander (Parts A + B) | 0 | 0 | 0 | 0 | 1 |  |  |  | 1
    Other (Parts A + B): number analyzed (Participants) | 14 | 16 | 37 | 85 | 46 | 0 | 0 | 0 | 198
    Other (Parts A + B) | 0 | 0 | 0 | 2 | 0 |  |  |  | 2
    Unknown (Parts A+B): number analyzed (Participants) | 14 | 16 | 37 | 85 | 0 | 0 | 0 | 0 | 152
    Unknown (Parts A+B) | 0 | 1 | 1 | 1 |  |  |  |  | 3
    Caucasian (Part C): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 50 | 51 | 51 | 152
    Caucasian (Part C) |  |  |  |  |  | 37 | 38 | 38 | 113
    Black (Part C): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 50 | 51 | 51 | 152
    Black (Part C) |  |  |  |  |  | 0 | 0 | 1 | 1
    Asian (Part C): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 50 | 51 | 51 | 152
    Asian (Part C) |  |  |  |  |  | 10 | 10 | 8 | 28
    Pacific Islander (Part C): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 50 | 51 | 51 | 152
    Pacific Islander (Part C) |  |  |  |  |  | 1 | 0 | 0 | 1
    Other (Part C): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 50 | 51 | 51 | 152
    Other (Part C) |  |  |  |  |  | 2 | 3 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Nonalcoholic Steatohepatitis (NASH) Patients With Treatment Emergent Adverse Events (TEAE)
Description: Number of Nonalcoholic steatohepatitis (NASH) patients with TEAEs
Time Frame: End of Treatment (EoT): For Parts A&B, EoT was Week 12 (Primary Outcome Measure). For Part C, EoT was Week 48 (Secondary Outcome Measure)
Population: Safety analysis set (SAS) is all subjects who received at least one dose of drug and had at least one post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Groups:
- LJN452 90 μg: 90 micrograms of Tropifexor (Parts A+B)
- LNJ452 200 μg: 200 micrograms of Tropifexor (Part C)
- Placebo Part C: Placebo (Part C)
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo A+B | LJN452 140 μg | LNJ452 200 μg | Placebo Part C
Number analyzed (Participants) | 13 | 17 | 37 | 85 | 46 | 50 | 51 | 51
Participants | 5 | 11 | 24 | 61 | 31 | 49 | 49 | 46

2. Primary Outcome: Change in Transaminase Levels (ALT)
Description: The alanine aminotransferase (ALT) test is a blood test that checks for liver damage. High levels of ALT may indicate liver damage. Normal range for ALT is typically 10 to 45 U/L or so (varies a little by age and gender). Elevation of these values indicate more liver inflammation/damage.
  ALT elevation is not unexpected in this patient population
  Dose relationship of tropifexor (LJN452) on ALT marker of hepatic inflammation in NASH from baseline to week 12
  Summary statistics of change in ALT from baseline to EOT by treatment
Time Frame: as for outcome 1
Population: Full analysis set (FAS): All subjects to whom study treatment had been assigned.
  Following the intent-to-treat (ITT) principle, subjects were analyzed according to the treatment they have been assigned to at randomization.
Measure: Mean (Standard Deviation); unit: IU/L
Groups:
- LJN452 60 μg: 60 micrograms of Tropifexor (Parts A + B)
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo A+B | LJN452 140 μg | LNJ452 200 μg | Placebo Part C
Number analyzed (Participants) | 14 | 16 | 37 | 85 | 46 | 50 | 51 | 51
IU/L | -16.7 (17.53) | -12.0 (35.99) | -17.3 (28.12) | -15.4 (30.32) | -8.1 (29.37) | -27.0 (30.24) | -28.7 (25.40) | -11.7 (61.64)
Statistical Analysis 1: Comparison: LJN452 10 μg vs Placebo A+B; 10 micrograms of Tropifexor vs placebo (Part A); Test type: Superiority — Repeated measures analysis: ALT (U/L) change from baseline up to EOT (Parts A + B) (Full analysis set); p = 0.362, ANCOVA; LS mean change = -15.9, 95% CI 2-sided [-31.2 to -0.6], Standard Error of Mean 7.76
Statistical Analysis 2: Comparison: LJN452 30 μg vs Placebo A+B; 30 micrograms of Tropifexor vs placebo (Part A); Test type: Superiority — Repeated measures analysis: ALT (U/L) change from baseline up to EOT (Parts A + B) (Full analysis set); p = 0.729, ANCOVA; LS mean change = -10.7, 95% CI 2-sided [-24.8 to 3.3], Standard Error of Mean 7.12
Statistical Analysis 3: Comparison: LJN452 60 μg vs Placebo A+B; 60 micrograms of Tropifexor vs placebo (Parts A + B); Test type: Superiority — Repeated measures analysis: ALT (U/L) change from baseline up to EOT (Parts A + B) (Full analysis set); p = 0.173, ANCOVA; Least Square Mean Change = -16.5, 95% CI 2-sided [-25.8 to -7.1], Standard Error of Mean 4.73
Statistical Analysis 4: Comparison: LJN452 90 μg vs Placebo A+B; 90 micrograms of Tropifexor vs placebo (Parts A + B); Test type: Superiority — Repeated measures analysis: ALT (U/L) change from baseline up to EOT (Parts A + B) (Full analysis set); p = 0.185, ANCOVA; Least Square Mean Change = -14.9, 95% CI 2-sided [-21.3 to -8.5], Standard Error of Mean 3.25
Statistical Analysis 5: Comparison: LJN452 140 μg vs Placebo Part C; 140 micrograms of Tropifexor (Part C) vs placebo; Test type: Superiority — Repeated measures analysis: ALT (U/L) change from baseline up to EOT (Part C) (Full analysis set); p = 0.020, ANCOVA; LS Mean Change = -31.6, 95% CI 2-sided [-46.9 to -16.3], Standard Error of Mean 7.71
Statistical Analysis 6: Comparison: LNJ452 200 μg vs Placebo Part C; 200 micrograms of Tropifexor vs placebo (Part C); Test type: Superiority — Repeated measures analysis: ALT (U/L) change from baseline up to EOT (Part C) (Full analysis set); p = 0.030, ANCOVA; LS Mean Change = -32.5, 95% CI 2-sided [-50.6 to -14.5], Standard Error of Mean 9.10
Statistical Analysis 7: Comparison: LJN452 10 μg vs Placebo A+B vs Placebo Part C; 10 micrograms of Tropifexor vs placebo (Parts A + B + C); Test type: Superiority — Repeated measures analysis: ALT (U/L) change from baseline to Week 12 (Parts A+B+C) Full analysis set (FAS); p = 0.456, ANCOVA; LS Mean change = -13.4, 95% CI 2-sided [-26.3 to -0.4], Standard Error of Mean 7.86
Statistical Analysis 8: Comparison: LJN452 30 μg vs Placebo A+B vs Placebo Part C; 30 micrograms of Tropifexor vs placebo (Parts A + B + C); Test type: Superiority — Repeated measures analysis: ALT (U/L) change from baseline to Week 12 (Parts A+B+C) Full analysis set (FAS); p = 0.966, ANCOVA; LS Mean change = -7.5, 95% CI 2-sided [-19.5 to 4.4], Standard Error of Mean 7.27
Statistical Analysis 9: Comparison: LJN452 60 μg vs Placebo A+B vs Placebo Part C; 60 micrograms of Tropifexor vs placebo (Parts A + B + C); Test type: Superiority — Repeated measures analysis: ALT (U/L) change from baseline to Week 12 (Parts A+B+C) Full analysis set (FAS); p = 0.275, ANCOVA; LS Mean change = -13.3, 95% CI 2-sided [-21.4 to -5.2], Standard Error of Mean 4.93
Statistical Analysis 10: Comparison: LJN452 90 μg vs Placebo A+B vs Placebo Part C; 90 micrograms of Tropifexor vs placebo (Parts A + B + C); Test type: Superiority — Repeated measures analysis: ALT (U/L) change from baseline to Week 12 (Parts A+B+C) Full analysis set (FAS); p = 0.304, ANCOVA; LS Mean change = -11.8, 95% CI 2-sided [-17.6 to -5.9], Standard Error of Mean 3.56
Statistical Analysis 11: Comparison: Placebo A+B vs LJN452 140 μg vs Placebo Part C; 140 micrograms of Tropifexor vs placebo (Parts A + B + C); Test type: Superiority — Repeated measures analysis: ALT (U/L) change from baseline up to EOT (Parts A + B) FAS; p = 0.057, ANCOVA; LS Mean change = -17.1, 95% CI 2-sided [-24.5 to -9.8], Standard Error of Mean 4.45
Statistical Analysis 12: Comparison: Placebo A+B vs LNJ452 200 μg vs Placebo Part C; 200 micrograms of Tropifexor vs placebo (Parts A + B + C); Test type: Superiority — Repeated measures analysis: ALT (U/L) change from baseline up to EOT (Parts A + B + C) FAS; p = 0.003, ANCOVA; LS Mean change = -23.0, 95% CI 2-sided [-30.5 to -15.6], Standard Error of Mean 4.49

3. Primary Outcome: Change in Aspartate Transaminase (AST)
Description: To determine the dose relationship of tropifexor (LJN452) on markers of hepatic inflammation (AST) in NASH from baseline to Week 12 The alanine aminotransferase (AST) test is a blood test that checks for liver damage. High levels of AST may indicate liver damage. Normal range for AST is typically 10 to 45 U/L or so (varies a little by age and gender). Elevation of these values indicate more liver inflammation/damage
  AST elevation is not unexpected in this patient population
  The aspartate aminotransferase (AST) test is a blood test that checks for liver damage. Higher levels indicate more possible liver damage
  Summary statistics of change in AST from baseline up to end of treatment (EOT)
Time Frame: as for outcome 1
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo A+B | LJN452 140 μg | LJN452 200 μg | Placebo Part C
Number analyzed (Participants) | 14 | 16 | 37 | 85 | 46 | 50 | 51 | 51
U/L | -11.3 (12.09) | -2.1 (29.62) | -10.2 (25.03) | -2.5 (24.60) | -7.1 (23.85) | -16.7 (23.36) | -13.3 (20.14) | -13.1 (29.00)
Statistical Analysis 1: Comparison: LJN452 10 μg vs Placebo A+B; 10 micrograms of Tropifexor vs placebo (Part A); Test type: Superiority — Repeated measures analysis: AST (U/L) change from baseline up to EOT (Full analysis set); p = 0.722, ANCOVA; LS Mean change = -9.9, 95% CI 2-sided [-22.9 to 3.0], Standard Error of Mean 6.56
Statistical Analysis 2: Comparison: LJN452 30 μg vs Placebo A+B; 30 micrograms of Tropifexor vs placebo (Part A); Test type: Superiority — Repeated measures analysis: AST (U/L) change from baseline up to EOT (Full analysis set); p = 0.468, ANCOVA; LS Mean change = -2.2, 95% CI 2-sided [-14.0 to 9.5], Standard Error of Mean 5.96
Statistical Analysis 3: Comparison: LJN452 60 μg vs Placebo A+B; 60 micrograms of Tropifexor vs placebo (Parts A+B); Test type: Superiority — Repeated measures analysis: AST (U/L) change from baseline up to EOT (Parts A+B) (Full analysis set); p = 0.774, ANCOVA; LS Mean change = -8.8, 95% CI 2-sided [-16.7 to -1.0], Standard Error of Mean 3.97
Statistical Analysis 4: Comparison: LJN452 90 μg vs Placebo A+B; 90 micrograms of Tropifexor vs placebo (Parts A+B); Test type: Superiority — Repeated measures analysis: AST (U/L) change from baseline up to EOT (Parts A+B) (Full analysis set); p = 0.136, ANCOVA; LS Mean change = -0.6, 95% CI 2-sided [-6.0 to 4.9], Standard Error of Mean 2.76
Statistical Analysis 5: Comparison: LJN452 140 μg vs Placebo Part C; 140 micrograms of Tropifexor vs placebo (Part C); Test type: Superiority — Repeated measures analysis: AST (U/L) change from baseline up to EOT (Part C) (Full analysis set); p = 0.145, ANCOVA; LS Mean change = -16.0, 95% CI 2-sided [-23.9 to -8.2], Standard Error of Mean 3.97
Statistical Analysis 6: Comparison: LJN452 200 μg vs Placebo Part C; 200 micrograms of Tropifexor vs placebo (Part C); Test type: Superiority — Repeated measures analysis: AST (U/L) change from baseline up to EOT (Part C) (Full analysis set); p = 0.236, ANCOVA; LS Mean change = -15.3, 95% CI 2-sided [-24.2 to -6.4], Standard Error of Mean 4.49
Statistical Analysis 7: Comparison: LJN452 10 μg vs Placebo A+B vs Placebo Part C; 10 micrograms of Tropifexor vs placebo (Parts A+B+ C); Test type: Superiority — Repeated measures analysis: AST (U/L) change from baseline up to EOT (Parts A+B+C) Full analysis set (FAS); p = 0.788, ANCOVA; LS Mean change = -7.1, 95% CI 2-sided [-18.7 to 4.4], Standard Error of Mean 7.00
Statistical Analysis 8: Comparison: LJN452 30 μg vs Placebo A+B vs Placebo Part C; 30 micrograms of Tropifexor vs placebo (Parts A+B+ C); Test type: Superiority — Repeated measures analysis: AST (U/L) change from baseline up to EOT (Parts A+B+C) Full analysis set (FAS); p = 0.413, ANCOVA; LS Mean change = 0.4, 95% CI 2-sided [-10.2 to 11.0], Standard Error of Mean 6.43
Statistical Analysis 9: Comparison: LJN452 60 μg vs Placebo A+B vs Placebo Part C; 60 micrograms of Tropifexor vs placebo (Parts A+B+ C); Test type: Superiority — Repeated measures analysis: AST (U/L) change from baseline up to EOT (Parts A+B+C) Full analysis set (FAS); p = 0.833, ANCOVA; LS Mean change = -6.2, 95% CI 2-sided [-13.4 to 1.0], Standard Error of Mean 4.38
Statistical Analysis 10: Comparison: LJN452 90 μg vs Placebo A+B vs Placebo Part C; 90 micrograms of Tropifexor vs placebo (Parts A+B+ C); Test type: Superiority — Repeated measures analysis: AST (U/L) change from baseline up to EOT (Parts A+B+C) Full analysis set (FAS); p = 0.068, ANCOVA; LS Mean change = 2.0, 95% CI 2-sided [-3.2 to 7.3], Standard Error of Mean 3.19
Statistical Analysis 11: Comparison: Placebo A+B vs LJN452 140 μg vs Placebo Part C; 140 micrograms of Tropifexor vs placebo (Parts A+B+ C); Test type: Superiority — Repeated measures analysis: AST (U/L) change from baseline up to EOT (Parts A+B+C) Full analysis set (FAS); p = 0.269, ANCOVA; LS Mean change = -0.1, 95% CI 2-sided [-6.6 to 6.5], Standard Error of Mean 3.98
Statistical Analysis 12: Comparison: Placebo A+B vs LJN452 200 μg vs Placebo Part C; 200 micrograms of Tropifexor vs placebo (Parts A+B+ C); Test type: Superiority — Repeated measures analysis: AST (U/L) change from baseline up to EOT (Parts A+B+C) Full analysis set (FAS); p = 0.777, ANCOVA; LS Mean change = -3.8, 95% CI 2-sided [-10.5 to 2.9], Standard Error of Mean 4.05

4. Primary Outcome: Change From Baseline in % of Fat in the Liver Assessed Using Magnetic Resonance Imaging (MRI)
Description: Repeated measures analysis: Relative change in percentage of fat in the liver assessed using MRI from baseline by visit up to EOT (Full analysis set)
Time Frame: as for outcome 1
Population: FAS
Measure: Mean (Standard Error); unit: percentage of fat in the liver
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo A+B | LJN452 140 μg | LJN452 200 μg | Placebo Part C
Number analyzed (Participants) | 14 | 16 | 37 | 85 | 46 | 50 | 51 | 51
percentage of fat in the liver | -7.48 (6.174) | -14.07 (5.661) | -15.04 (3.754) | -12.34 (2.482) | -6.19 (3.381) | -31.25 (5.228) | -39.54 (4.968) | -3.58 (4.718)
Statistical Analysis 1: Comparison: LJN452 10 μg vs Placebo A+B; 10 microgramsof Tropifexor - Change in percentage of fat in the liver Part A; Test type: Superiority — ANCOVA: Relative change in percentage of fat in the liver from baseline to Week 12; p = 0.853, ANCOVA; LS Mean change = -7.48, 95% CI 2-sided [-19.66 to 4.70], Standard Error of Mean 6.174
Statistical Analysis 2: Comparison: LJN452 30 μg vs Placebo A+B; 30 micrograms of Tropifexor - Change in percentage of fat in the liver Part A; Test type: Superiority — ANCOVA: Relative change in percentage of fat in the liver from baseline to Week 12; p = 0.232, ANCOVA; LS Mean change = -14.07, 95% CI 2-sided [-25.24 to -2.91], Standard Error of Mean 5.661
Statistical Analysis 3: Comparison: LJN452 60 μg vs Placebo A+B; 60 micrograms of Tropifexor - Change in percentage of fat in the liver Parts A+B; Test type: Superiority — ANCOVA: Relative change in percentage of fat in the liver from baseline to Week 12; p = 0.077, ANCOVA; LS Mean change = -15.04, 95% CI 2-sided [-22.45 to -7.64], Standard Error of Mean 3.754
Statistical Analysis 4: Comparison: LJN452 90 μg vs Placebo A+B; 90 micrograms of Tropifexor - Change in percentage of fat in the liver Parts A+B; Test type: Superiority — ANCOVA: Relative change in percentage of fat in the liver from baseline; p = 0.141, ANCOVA; LS Mean change = -12.34, 95% CI 2-sided [-17.23 to -7.44], Standard Error of Mean 2.482
Statistical Analysis 5: Comparison: LJN452 140 μg vs Placebo Part C; 140 micrograms of Tropifexor - Change in percentage of fat in the liver Part C; Test type: Superiority — ANCOVA: Relative change in percentage of fat in the liver from baseline to Week 12; p < 0.001, ANCOVA; LS Mean change = -31.25, 95% CI 2-sided [-41.58 to -20.92], Standard Error of Mean 5.228
Statistical Analysis 6: Comparison: LJN452 200 μg vs Placebo Part C; 200 micrograms of Tropifexor - Change in percentage of fat in the liver Part C; Test type: Superiority — ANCOVA: Relative change in percentage of fat in the liver from baseline to Week 12 (Parts A+B+C); p < 0.001, ANCOVA; LS Mean change = -39.54, 95% CI 2-sided [-49.37 to -29.71], Standard Error of Mean 4.968
Statistical Analysis 7: Comparison: LJN452 10 μg vs Placebo A+B vs Placebo Part C; 10 micrograms of Tropifexor - Change in percentage of fat in the liver Parts A+B+C; Test type: Superiority — ANCOVA: Relative change in percentage of fat in the liver from baseline to Week 12 (Parts A+B+C); p = 0.872, ANCOVA; LS Mean change = -8.09, 95% CI 2-sided [-19.06 to 2.88], Standard Error of Mean 6.650
Statistical Analysis 8: Comparison: LJN452 30 μg vs Placebo A+B vs Placebo Part C; 30 micrograms of Tropifexor - Change in percentage of fat in the liver Parts A+B+C; Test type: Superiority — ANCOVA: Relative change in percentage of fat in the liver from baseline to Week 12 (Parts A+B+C); p = 0.465, ANCOVA; LS Mean change = -14.14, 95% CI 2-sided [-24.36 to -3.91], Standard Error of Mean 6.198
Statistical Analysis 9: Comparison: LJN452 60 μg vs Placebo A+B vs Placebo Part C; 60 micrograms of Tropifexor - Change in percentage of fat in the liver Parts A+B+C; Test type: Superiority — ANCOVA: Relative change in percentage of fat in the liver from baseline to Week 12 (Parts A+B+C); p = 0.228, ANCOVA; LS Mean change = -15.02, 95% CI 2-sided [-21.75 to -8.29], Standard Error of Mean 4.078
Statistical Analysis 10: Comparison: LJN452 90 μg vs Placebo A+B vs Placebo Part C; 90 micrograms - Change in percentage of fat in the liver Parts A+B+C; Test type: Superiority — ANCOVA: Relative change in percentage of fat in the liver from baseline to Week 12 (Parts A+B+C); p = 0.370, ANCOVA; LS Mean change = -12.56, 95% CI 2-sided [-17.04 to -8.08], Standard Error of Mean 2.717
Statistical Analysis 11: Comparison: Placebo A+B vs LJN452 140 μg vs Placebo Part C; 140 micrograms - Change in percentage of fat in the liver Parts A+B+C; Test type: Superiority — ANCOVA: Relative change in percentage of fat in the liver from baseline to Week 12 (Parts A+B+C); p = 0.029, ANCOVA; LS Mean change = -18.71, 95% CI 2-sided [-24.51 to -12.91], Standard Error of Mean 3.517
Statistical Analysis 12: Comparison: Placebo A+B vs LJN452 200 μg vs Placebo Part C; 200 micrograms of Tropifexor - Change in percentage of fat in the liver Parts A+B+C; Test type: Superiority — ANCOVA: Relative change in percentage of fat in the liver from baseline to Week 12 (Parts A+B+C); p < 0.001, ANCOVA; LS Mean change = -34.38, 95% CI 2-sided [-40.13 to -28.64], Standard Error of Mean 3.482

5. Secondary Outcome: Change From Baseline in Weight
Description: Repeated measures for LS mean change in weight after 12 weeks of treatment
Time Frame: 48 weeks
Population: FAS
Measure: Mean (Standard Error); unit: kg
Groups:
- LJN452 30 μg: 30 micrograms of Tropifexor (Part A) vs placebo
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo A+B | LJN452 140 μg | LJN452 200 μg | Placebo Part C
Number analyzed (Participants) | 14 | 16 | 36 | 84 | 46 | 50 | 51 | 51
kg | -1.79 (0.608) | -0.78 (0.567) | -1.05 (0.377) | -1.15 (0.253) | 0.00 (0.338) | -5.10 (0.988) | -5.89 (1.002) | -2.48 (0.915)
Statistical Analysis 1: Comparison: LJN452 10 μg vs Placebo A+B; 10 micrograms of Tropifexor (Part A) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in weight from baseline to EOT (Parts A + B) (Full analysis set); p = 0.010, Mixed Models Analysis; LS Mean change = -1.79, 95% CI 2-sided [-2.99 to 0.59], Standard Error of Mean 0.608
Statistical Analysis 2: Comparison: LJN452 30 μg vs Placebo A+B; 30 micrograms of Tropifexor (Part A) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in weight from baseline to EOT (Parts A + B) (Full analysis set); p = 0.237, Mixed Models Analysis; LS Mean change = -0.78, 95% CI 2-sided [-1.90 to 0.34], Standard Error of Mean 0.567
Statistical Analysis 3: Comparison: LJN452 60 μg vs Placebo A+B; 60 micrograms of Tropifexor (Parts A + B) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in weight from baseline to EOT (Parts A + B) (Full analysis set); p = 0.037, Mixed Models Analysis; LS Mean change = -1.05, 95% CI 2-sided [-1.80 to 0.31], Standard Error of Mean 0.377
Statistical Analysis 4: Comparison: LJN452 90 μg vs Placebo A+B; 90 micrograms of Tropifexor (Parts A + B) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in weight from baseline to EOT (Parts A + B) (Full analysis set); p = 0.007, Mixed Models Analysis; LS Mean change = -1.15, 95% CI 2-sided [-1.65 to 0.65], Standard Error of Mean 0.253
Statistical Analysis 5: Comparison: LJN452 140 μg vs Placebo Part C; 140 micrograms of Tropifexor (Part C) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in weight from baseline to EOT (Parts C) (Full analysis set); p = 0.053, Mixed Models Analysis; LS Mean change = -5.10, 95% CI 2-sided [-7.05 to -3.14], Standard Error of Mean 0.988
Statistical Analysis 6: Comparison: LJN452 200 μg vs Placebo Part C; 200 micrograms of Tropifexor (Part C) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in weight from baseline to EOT (Parts C) (Full analysis set); p = 0.013, Mixed Models Analysis; LS Mean change = -5.89, 95% CI 2-sided [-7.87 to -3.91], Standard Error of Mean 1.002

6. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Repeated measures for the LS mean change in BMI after 12 weeks of treatment. Body mass index (BMI) is a measure of body fat based on height and weight
Time Frame: 12 weeks
Population: FAS
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo A+B | LJN452 140 μg | LJN452 200 μg | Placebo Part C
Number analyzed (Participants) | 14 | 16 | 37 | 84 | 46 | 50 | 51 | 51
kg/m2 | -0.64 (0.208) | -0.29 (0.194) | -0.35 (0.129) | -0.42 (0.087) | 0.02 (0.116) | -1.88 (0.322) | -2.11 (0.327) | -0.80 (0.299)
Statistical Analysis 1: Comparison: LJN452 10 μg vs Placebo A+B; 10 micrograms of Tropifexor (Part A) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in BMI from baseline to EOT (Full analysis set); p = 0.006, Mixed Models Analysis; LS Mean change = -0.64, 95% CI 2-sided [-1.05 to 0.23], Standard Error of Mean 0.208
Statistical Analysis 2: Comparison: LJN452 30 μg vs Placebo A+B; 30 micrograms of Tropifexor (Part A) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in BMI from baseline to EOT (Full analysis set); p = 0.177, Mixed Models Analysis; LS Mean change = -0.29, 95% CI 2-sided [-0.67 to 0.09], Standard Error of Mean 0.194
Statistical Analysis 3: Comparison: LJN452 60 μg vs Placebo A+B; 60 micrograms of Tropifexor (Parts A + B) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in BMI from baseline to EOT (Parts C) (Full analysis set); p = 0.032, Mixed Models Analysis; LS Mean change = -0.35, 95% CI 2-sided [-0.61 to 0.10], Standard Error of Mean 0.129
Statistical Analysis 4: Comparison: LJN452 90 μg vs Placebo A+B; 90 micrograms of Tropifexor (Parts A + B) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in BMI from baseline to EOT (Full analysis set); p = 0.003, Mixed Models Analysis; LS Mean change = -0.42, 95% CI 2-sided [-0.59 to 0.25], Standard Error of Mean 0.087
Statistical Analysis 5: Comparison: LJN452 140 μg vs Placebo Part C; 140 micrograms of Tropifexor (Part C) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in BMI from baseline to EOT (Full analysis set); p = 0.015, Mixed Models Analysis; LS Mean change = -1.88, 95% CI 2-sided [-2.51 to -1.24], Standard Error of Mean 0.322
Statistical Analysis 6: Comparison: LJN452 200 μg vs Placebo Part C; 200 micrograms of Tropifexor (Part C) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in BMI from baseline to EOT (Parts C) (Full analysis set); p = 0.004, Mixed Models Analysis; LS Mean change = -2.11, 95% CI 2-sided [-2.75 to -1.46], Standard Error of Mean 0.327

7. Secondary Outcome: Change From Baseline in Waist to Hip (WTH) Ratio
Description: The LS mean change in waist to hip ratio after 12 weeks of treatment
Time Frame: 12 weeks
Population: FAS
Measure: Mean (Standard Error); unit: ratio
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo A+B | LJN452 140 μg | LJN452 200 μg | Placebo Part C
Number analyzed (Participants) | 13 | 15 | 37 | 84 | 46 | 49 | 37 | 51
ratio | -0.01 (0.009) | 0.00 (0.008) | -0.01 (0.005) | 0.00 (0.004) | 0.00 (0.005) | 0.00 (0.008) | -0.01 (0.007) | -0.02 (0.007)
Statistical Analysis 1: Comparison: LJN452 10 μg vs Placebo A+B; 10 micrograms of Tropifexor (Part A) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in WTH ratio from baseline to EOT (Parts A+B) (Full analysis set); p = 0.530, Mixed Models Analysis; LS Mean change = -0.01, 95% CI 2-sided [-0.03 to 0.01], Standard Error of Mean 0.009
Statistical Analysis 2: Comparison: LJN452 30 μg vs Placebo A+B; 30 micrograms of Tropifexor (Part A) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in WTH ratio from baseline to EOT (Parts A+B) (Full analysis set); p = 0.857, Mixed Models Analysis; LS Mean change = 0.00, 95% CI 2-sided [-0.02 to 0.01], Standard Error of Mean 0.008
Statistical Analysis 3: Comparison: LJN452 60 μg vs Placebo A+B; 60 micrograms of Tropifexor (Part A) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in WTH ratio from baseline to EOT (Parts A+B) (Full analysis set); p = 0.262, Mixed Models Analysis; LS Mean change = -0.01, 95% CI 2-sided [-0.02 to 0.00], Standard Error of Mean 0.005
Statistical Analysis 4: Comparison: LJN452 90 μg vs Placebo A+B; 90 micrograms of Tropifexor (Parts A + B) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in WTH ratio from baseline to EOT (Parts A+B) (Full analysis set); p = 0.323, Mixed Models Analysis; LS Mean change = 0.00, 95% CI 2-sided [0.00 to 0.01], Standard Error of Mean 0.004
Statistical Analysis 5: Comparison: LJN452 140 μg vs Placebo Part C; 140 micrograms of Tropifexor (Part C) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in WTH ratio from baseline to EOT (Part C) (Full analysis set); p = 0.100, Mixed Models Analysis; LS Mean change = 0.01, 95% CI 2-sided [-0.02 to 0.01], Standard Error of Mean 0.008
Statistical Analysis 6: Comparison: LJN452 200 μg vs Placebo Part C; 200 micrograms of Tropifexor (Part C) vs Placebo; Test type: Superiority — Repeated measures analysis: Change in WTH ratio from baseline to EOT (Part C) (Full analysis set); p = 0.693, Mixed Models Analysis; LS Mean change = -0.01, 95% CI 2-sided [-0.03 to 0.00], Standard Error of Mean 0.007

8. Secondary Outcome: Change From Baseline in Biomarker FGF19
Description: Dose-response relationship of tropifexor (LJN452) on FGF19 over time, a marker of FXR target engagement in the gut.
  ANCOVA: Ratio of FGF19 (pg/mL) post-dose to pre-dose at Week 6
  Value at 6 weeks minus value at baseline
Time Frame: baseline, week 6
Population: FAS
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo A+B | LJN452 140 μg | LJN452 200 μg | Placebo Part C
Number analyzed (Participants) | 14 | 15 | 34 | 78 | 42 | 47 | 42 | 42
pg/mL | 1.45 [0.93 to 2.26] | 1.53 [1.00 to 2.35] | 3.82 [2.88 to 5.09] | 5.78 [4.78 to 6.98] | 1.33 [1.03 to 1.73] | 1.97 [1.48 to 2.62] | 2.23 [1.65 to 3.01] | 1.22 [0.92 to 1.61]

9. Secondary Outcome: Change From Baseline in Biomarker C4
Description: Dose-response relationship of LJN452 on C4, a marker of hepatic target engagement at 4 hours post dose
  C4 (ng/mL): Summary statistics by treatment and visit
Time Frame: Week 6, 4 hours post dose
Population: FAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo A+B | LJN452 140 μg | LJN452 200 μg | Placebo Part C
Number analyzed (Participants) | 14 | 15 | 37 | 85 | 46 | 47 | 42 | 51
ng/mL | 38.82 (25.765) | 32.75 (23.360) | 28.38 (13.394) | 40.19 (31.356) | 47.70 (25.524) | 14.97 (20.232) | 8.54 (9.583) | 38.40 (24.552)

10. Secondary Outcome: Change From Baseline on Markers of Liver Fibrosis, Fibroscan
Description: Dose-response relationship of tropifexor (LJN452) on markers of liver fibrosis commonly available such as Fibroscan®
  Liver stiffness (kPa): Summary statistics by treatment and visit
  FibroScan is a specialized ultrasound machine for measuring fibrosis (scarring) in the liver
  Scores range from 0-4 with zero being no liver scarring and 4 being advanced liver scarring (cirrhosis)
Time Frame: End of Treatment (EoT): For Parts A&B, EoT was Week 12. For Part C, EoT was Week 48
Population: FAS
Measure: Mean (Standard Deviation); unit: scores
Groups:
- Placebo (Part C): Placebo (Part C)
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo A+B | LJN452 140 μg | LJN452 200 μg | Placebo (Part C)
Number analyzed (Participants) | 14 | 16 | 37 | 85 | 46 | 46 | 42 | 51
scores | 10.94 (5.314) | 10.40 (7.663) | 9.90 (4.095) | 9.00 (4.152) | 9.30 (4.676) | 11.29 (3.677) | 12.03 (4.804) | 11.26 (4.027)

11. Secondary Outcome: Change From Baseline on Markers of Liver Fibrosis Panel (ELF) Score
Description: ANCOVA: LS Mean Change in Enhanced liver fibrosis panel (ELF) score from baseline by visit up to EOT.
  The total ELF score reference range calculated non-parametrically is 6.72 (90% CI 6.58-6.84) to 9.79 (90% CI 9.45-10.01); Journal of Hepatology 2013 vol. 59 j 236-242.
  Enhanced liver fibrosis Test (ELF) panel: the following was assessed: hyaluronic acid (HA), tissue inhibitor of metalloproteinases (TIMP-1), and amino-terminal pro-peptide of procollagen type III (PIIINP).
  The Enhanced Liver Fibrosis score is a linear combination of TIMP-1, PIIINP, and HA with the following formula: ELF score = 2.494+0.846 x ln(HA) + 0.735 x ln (PIIINP) + 0.391 x ln (TIMP-1).
Time Frame: End of Treatment (EoT): For Parts A&B, EoT was Week 12. For Part C, EoT was Week 48
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Groups:
- LJN452 30 μg: 30 micrograms of Tropifexor (Parts A + B)
- LJN452 140 μg: 140 micrograms of Tropifexor (Part C) vs placebo
- Placebo Part C: (Part C)
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo A+B | LJN452 140 μg | LJN452 200 μg | Placebo Part C
Number analyzed (Participants) | 14 | 16 | 34 | 78 | 46 | 47 | 42 | 51
scores on a scale | 0.05 (0.158) | 0.00 (0.146) | -0.19 (0.097) | 0.20 (0.064) | 0.08 (0.087) | -0.34 (0.132) | -0.24 (0.122) | -0.08 (0.115)

12. Secondary Outcome: Change From Baseline on Markers of Liver Fibrosis, Fibrotest (Parts A+B)
Description: Fibrosis biomarker test, originally called Fibrotest®/ Fibrosure®, is combines α2-macroglobulin (a2m), apolipoprotein A1 (aA1), total bilirubin (BIL), haptoglobin (h), GGT, and ALT. The coefficient for the score is calculated as: z = 4.467 x log(a2m) - 1.357 x log(h) + 1.017 x log(GGT) + 0.0281 x Age + 1.737 x log(BIL) - 1.184 x (aA1) + 0.301 x Gender - 5.54 where Gender = 1 for male and Gender = 0 for female. The score is then: 1/(1+e^-z).
  Calculated scores range from 0.00 (no fibrosis) to 1.00 (severe fibrosis or cirrhosis) (See Part C in separate outcomes that follows)
Time Frame: End of Treatment (EoT):12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: scores
Groups:
- Placebo (A+B): Placebo (Parts A+B)
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo (A+B)
Number analyzed (Participants) | 14 | 16 | 37 | 85 | 46
scores | -0.23 (0.284) | -1.49 (0.852) | -1.44 (1.080) | -1.34 (1.222) | -1.23 (1.088)

13. Secondary Outcome: Change From Baseline on Markers of Liver Fibrosis, Fibrotest, (Part C)
Description: Fibrosis biomarker test, originally called Fibrotest®/ Fibrosure®, is combines α2-macroglobulin (a2m), apolipoprotein A1 (aA1), total bilirubin (BIL), haptoglobin (h), GGT, and ALT. The coefficient for the score is calculated as: z = 4.467 x log(a2m) - 1.357 x log(h) + 1.017 x log(GGT) + 0.0281 x Age + 1.737 x log(BIL) - 1.184 x (aA1) + 0.301 x Gender - 5.54 where Gender = 1 for male and Gender = 0 for female. The score is then: 1/(1+e^-z).
  Calculated scores range from 0.00 (no fibrosis) to 1.00 (severe fibrosis or cirrhosis)
Time Frame: End of Treatment (EoT) was 48 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores
Arm/Group | LJN452 140 μg | LJN452 200 μg | Placebo A+B
Number analyzed (Participants) | 34 | 28 | 37
scores | -0.42 (0.131) | -0.44 (0.135) | -0.17 (0.119)

14. Secondary Outcome: Change From Baseline on Gamma-glutamyl Transferase (GGT)
Description: Summary statistics of change in GGT (IU/L) from baseline by visit up to EoT
Time Frame: EoT for Parts A+B=12 weeks; EoT for Part C = 48 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: IU/L
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo A+B | LJN452 140 μg | LJN452 200 μg | Placebo C
Number analyzed (Participants) | 14 | 15 | 37 | 84 | 78 | 51 | 42 | 36
IU/L | 1.6 (10.93) | -29.9 (10.11) | -34.2 (6.70) | -45.7 (4.52) | -5.0 (6.10) | -35.2 (11.58) | -29.9 (11.65) | 9.0 (10.72)

15. Secondary Outcome: Change From Baseline on Fasting Lipid Profile
Description: Repeated measures analysis: LS geometric mean ratio of fasting lipids to baseline by visit up to EOT
Time Frame: End of Treatment (EoT): For Parts A&B, EoT was Week 12. For Part C, EoT was Week 48
Population: FAS
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo A+B | LJN452 140 μg | LJN452 200 μg | Placebo Part C
Number analyzed (Participants) | 14 | 16 | 37 | 50 | 46 | 46 | 42 | 37
mmol/L
  Cholesterol | 0.949 [0.888 to 1.014] | 1.003 [0.945 to 1.065] | 1.029 [0.989 to 1.070] | 1.029 [1.002 to 1.057] | 0.956 [0.923 to 0.991] | 1.032 [0.975 to 1.093] | 1.071 [1.012 to 1.133] | 0.977 [0.928 to 1.029]
  Triglycerides | 0.920 [0.766 to 1.091] | 0.919 [0.789 to 1.071] | 0.960 [0.868 to 1.062] | 1.048 [0.978 to 1.123] | 0.991 [0.904 to 1.085] | 1.070 [0.934 to 1.226] | 1.068 [0.936 to 1.219] | 0.883 [0.782 to 0.998]
  LDL Cholesterol | 0.923 [0.834 to 1.020] | 1.044 [0.953 to 1.142] | 1.092 [1.029 to 1.159] | 1.104 [1.060 to 1.150] | 0.943 [0.893 to 0.995] | 1.056 [0.972 to 1.147] | 1.200 [1.106 to 1.302] | 0.973 [0.903 to 1.049]
  HDL Cholesterol | 1.019 [0.946 to 1.096] | 1.001 [0.937 to 1.069] | 0.961 [0.920 to 1.004] | 0.897 [0.870 to 0.924] | 0.959 [0.922 to 0.998] | 0.855 [0.800 to 0.913] | 0.824 [0.772 to 0.879] | 1.033 [0.973 to 1.096]
  LDL/HDL Ratio | 0.921 [0.810 to 1.047] | 1.058 [0.942 to 1.188] | 1.139 [1.055 to 1.229] | 1.227 [1.165 to 1.293] | 0.980 [0.915 to 1.051] | 1.252 [1.128 to 1.390] | 1.478 [1.332 to 1.639] | 0.947 [0.862 to 1.041]
  Free Glycerol | 1.0563 [0.8722 to 1.2793] | 0.9376 [0.7859 to 1.1185] | 0.9128 [0.8112 to 1.0272] | 0.9915 [0.9151 to 1.0743] | 0.9604 [0.8641 to 1.0674] | 1.1115 [0.9721 to 1.2709] | 0.9808 [0.8571 to 1.1223] | 0.9846 [0.8722 to 1.11116]
  Free Fatty Acid | 1.082 [0.897 to 1.305] | 0.864 [0.726 to 1.028] | 0.929 [0.827 to 1.043] | 0.947 [0.874 to 1.025] | 0.936 [0.844 to 1.038] | 1.072 [0.951 to 1.208] | 0.887 [0.785 to 1.002] | 0.977 [0.928 to 1.029]

16. Secondary Outcome: Itch Based on a Visual Analog Scale (VAS) Rating Scale
Description: Repeated measures analysis: Change in VAS for Itch from baseline by visit up to EoT
  VAS score 0 = no disease; and 9 is severely advanced disease
Time Frame: EoT for Parts A+B=12 weeks; EoT for Part C = 48 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores
Groups:
- LJN452 60 μg: 60 micrograms of Tropifexor (Parts A + B) vs placebo
- Placebo A+B: Placebo for parts A + B
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | Placebo A+B | LJN452 140 μg | LJN452 200 μg | Placebo Part C
Number analyzed (Participants) | 14 | 16 | 36 | 78 | 39 | 47 | 42 | 37
scores | -0.3 (0.48) | 0.2 (0.43) | 0.4 (0.28) | 0.1 (0.19) | 0.6 (0.27) | 0.6 (0.37) | 1.1 (0.35) | 0.3 (0.33)

17. Secondary Outcome: Pre-dose Trough Concentration (Ctrough) of LJN452
Description: Pre-dose Trough Concentration (Ctrough) of tropifexor (LJN452)
Time Frame: In Parts A and B, LJN452 Ctrough was measured on Study Days 7, 14, 28, 42, 56, and 84. In Part C LJN452 Ctrough was measured on Study Days 42, 84, 168, 280 and 336
Population: FAS
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- LJN452 10 μg: 10 micrograms of Tropifexor (Parts A + B)
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | LJN452 140 μg | LJN452 200 μg
Number analyzed (Participants) | 14 | 16 | 37 | 85 | 37 | 51
ng/mL
  Profile day 7: number analyzed (Participants) | 14 | 16 | 37 | 85 | 0 | 0
  Profile day 7 | 0.142 (0.119) | 0.355 (0.194) | 0.638 (0.453) | 1.215 (0.593) |  |
  Profile day 14: number analyzed (Participants) | 14 | 16 | 37 | 85 | 0 | 0
  Profile day 14 | 0.216 (0.127) | 0.505 (0.328) | 0.626 (0.281) | 1.115 (0.693) |  |
  Profile day 28: number analyzed (Participants) | 14 | 16 | 37 | 85 | 0 | 0
  Profile day 28 | 0.118 (0.087) | 0.411 (0.250) | 0.639 (0.265) | 1.027 (0.700) |  |
  Profile day 42 | 0.161 (0.094) | 0.382 (0.150) | 0.647 (0.344) | 1.032 (0.661) | 2.821 (1.659) | 3.533 (2.356)
  Profile day 56: number analyzed (Participants) | 14 | 16 | 37 | 85 | 0 | 0
  Profile day 56 | 0.168 (0.088) | 0.474 (0.273) | 0.637 (0.278) | 1.041 (0.701) |  |
  Profile day 84 | 0.118 (0.080) | 0.366 (0.147) | 0.530 (0.357) | 1.095 (0.653) | 1.685 (0.874) | 2.286 (1.259)
  Profile day 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 37 | 51
  Profile day 168 |  |  |  |  | 1.889 (1.340) | 2.146 (1.383)
  Profile day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 37 | 51
  Profile day 280 |  |  |  |  | 2.129 (1.257) | 1.990 (1.053)
  Profile day 336: number analyzed (Participants) | 0 | 0 | 0 | 0 | 37 | 51
  Profile day 336 |  |  |  |  | 1.444 (1.077) | 1.979 (1.153)

18. Secondary Outcome: C2h (Steady-state Drug Levels 2 Hours Postdose) of LJN452
Description: Summary C2h of tropifexor (LJN452)
Time Frame: Days 7 and 14 (10 and 30μg LJN452 C2h was not measured day 14)
Population: FAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg
Number analyzed (Participants) | 14 | 16 | 37 | 85
ng/mL
  Profile day 7 | 0.190 (0.143) | 0.702 (0.399) | 1.228 (0.598) | 2.193 (1.003)
  Profile day 14: number analyzed (Participants) | 0 | 0 | 37 | 85
  Profile day 14 |  |  | 1.344 (0.727) | 2.001 (1.053)

19. Secondary Outcome: Biopsy-based Response at Week 48 Compared to Baseline: At Least One Point Improvement in Fibrosis (NASH CRN Staging) Without Worsening of Steatohepatitis (Part C) - Total Score
Description: Number of patients who have at least one point improvement in fibrosis (NASH CRN staging) without worsening of steatohepatitis (total score)
Time Frame: EoT (Week 48)
Population: Full analysis set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | LJN452 140 μg | LNJ452 200 μg | Placebo C
Number analyzed (Participants) | 39 | 35 | 42
Participants | 11 | 11 | 12
Statistical Analysis 1: Comparison: LJN452 140 μg vs Placebo C; At least one point improvement in fibrosis (NASH CRN staging) without worsening of steatohepatitis (total score); Test type: Superiority; p = 1.0000, Mixed Models Analysis; Risk Difference (RD) = 0.004, 95% CI 2-sided [-0.214 to 0.223]
Statistical Analysis 2: Comparison: LNJ452 200 μg vs Placebo C; At least one point improvement in fibrosis (NASH CRN staging) without worsening of steatohepatitis (total score); Test type: Superiority; p = 0.8074, Mixed Models Analysis; Risk Difference (RD) = 0.029, 95% CI 2-sided [-0.196 to 0.251]

20. Secondary Outcome: Biopsy-based Response at Week 48 Compared to Baseline: At Least One Point Improvement in Fibrosis (NASH CRN Staging) Without Worsening - FDA
Description: Number of patients who have at least one point improvement in fibrosis (NASH CRN staging) without worsening of steatohepatitis (FDA)
Time Frame: EoT (Week 48)
Population: Full analysis set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | LJN452 140 μg | LNJ452 200 μg | Placebo A+B
Number analyzed (Participants) | 38 | 35 | 42
Participants | 11 | 11 | 11
Statistical Analysis 1: Comparison: LJN452 140 μg vs Placebo A+B; At least one point improvement in fibrosis (NASH CRN staging) without worsening of steatohepatitis (FDA); Test type: Superiority; p = 0.8070, Mixed Models Analysis; Risk Difference (RD) = 0.028, 95% CI 2-sided [-0.191 to 0.246]
Statistical Analysis 2: Comparison: LNJ452 200 μg vs Placebo A+B; At least one point improvement in fibrosis (NASH CRN staging) without worsening of steatohepatitis (FDA); Test type: Superiority; p = 0.6233, Mixed Models Analysis; Risk Difference (RD) = 0.052, 95% CI 2-sided [-0.173 to 0.273]

21. Secondary Outcome: Biopsy-based Response at Week 48 Compared to Baseline: At Least One Point Improvement in Fibrosis (NASH CRN Staging) Without Worsening - EMA
Description: Number of patients who have at least one point improvement in fibrosis (NASH CRN staging) without worsening of steatohepatitis (EMA)
Time Frame: EoT (Week 48)
Population: Full analysis set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | LJN452 140 μg | LNJ452 200 μg | Placebo A+B
Number analyzed (Participants) | 38 | 35 | 42
Participants | 11 | 11 | 12
Statistical Analysis 1: Comparison: LJN452 140 μg vs Placebo A+B; At least one point improvement in fibrosis (NASH CRN staging) without worsening of steatohepatitis (EMA); Test type: Superiority; p = 1.0000, Mixed Models Analysis; Risk Difference (RD) = 0.004, 95% CI 2-sided [-0.214 to 0.233]
Statistical Analysis 2: Comparison: LNJ452 200 μg vs Placebo A+B; At least one point improvement in fibrosis (NASH CRN staging) without worsening of steatohepatitis (EMA); Test type: Superiority; p = 0.8074, Mixed Models Analysis; Risk Difference (RD) = 0.029, 95% CI 2-sided [-0.196 to 0.251]

22. Secondary Outcome: Biopsy-based Response at Week 48 Compared to Baseline: Difference Between Treatment Groups (Part C) - Resolution of Steatohepatitis (Diagnostic Category)
Description: Resolution of steatohepatitis (diagnostic category) without worsening of fibrosis (NASH CRN staging)
Time Frame: EoT (Week 48)
Population: Full analysis set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | LJN452 140 μg | LNJ452 200 μg | Placebo A+B
Number analyzed (Participants) | 38 | 35 | 42
Participants | 4 | 7 | 3
Statistical Analysis 1: Comparison: LJN452 140 μg vs Placebo A+B; Resolution of steatohepatitis (diagnostic category) without worsening of fibrosis (NASH CRN staging); Test type: Superiority; p = 0.7028, Mixed Models Analysis; Risk Difference (RD) = 0.034, 95% CI 2-sided [-0.184 to 0.252]
Statistical Analysis 2: Comparison: LNJ452 200 μg vs Placebo A+B; Resolution of steatohepatitis (diagnostic category) without worsening of fibrosis (NASH CRN staging); Test type: Superiority; p = 0.1713, Mixed Models Analysis; Risk Difference (RD) = 0.129, 95% CI 2-sided [-0.098 to 0.345]

23. Secondary Outcome: Biopsy-based Response at Week 48 Compared to Baseline: Difference Between Treatment Groups (Part C) - Resolution of Steatohepatitis (FDA, EMA)
Description: Resolution of steatohepatitis (diagnostic category) without worsening of fibrosis (NASH CRN staging)
Time Frame: EoT (Week 48)
Population: Full analysis set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | LJN452 140 μg | LNJ452 200 μg | Placebo A+B
Number analyzed (Participants) | 38 | 35 | 42
Participants | 0 | 2 | 0
Statistical Analysis 1: Comparison: LNJ452 200 μg vs Placebo A+B; Resolution of steatohepatitis (FDA, EMA) without worsening of fibrosis (NASH CRN staging); Test type: Superiority; p = 0.2033, Mixed Models Analysis; Risk Difference (RD) = 0.057, 95% CI 2-sided [-0.168 to 0.278]

ADVERSE EVENTS:
Time Frame: To End of Treatment (EoT): For Parts A&B, EoT was Week 12; For Part C, EoT was Week 48
Description: AEs are any untoward sign or symptom that occurred during the study treatment period
  350 patients were randomized. One patient was treated at 2 sites, so 351 enrolled may appearr in some places.
Groups:
- LJN452 10 μg: LJN452 10 mcg (Part A)
- LJN452 60 μg: LJN452 60 mcg (Parts A+B)
- LJN452 140 μg: LJN452 140 mcg (Part C)
- LJN452 200 μg: LJN452 200 mcg (Part C)
- Placebo: Placebo A+B+C
- Total: Total
Arm/Group | LJN452 10 μg | LJN452 30 μg | LJN452 60 μg | LJN452 90 μg | LJN452 140 μg | LJN452 200 μg | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/17 | 0/37 | 0/85 | 0/50 | 0/51 | 0/97 | 0/350
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/17 | 0/37 | 4/85 | 5/50 | 3/51 | 6/97 | 18/350
Other Adverse Events (participants affected / at risk) | 5/13 | 11/17 | 16/37 | 50/85 | 43/50 | 45/51 | 63/97 | 233/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LJN452 10 μg (N=13) | LJN452 30 μg (N=17) | LJN452 60 μg (N=37) | LJN452 90 μg (N=85) | LJN452 140 μg (N=50) | LJN452 200 μg (N=51) | Placebo (N=97) | Total (N=350)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Device dislocation (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Endometrial thickening (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LJN452 10 μg (N=13) | LJN452 30 μg (N=17) | LJN452 60 μg (N=37) | LJN452 90 μg (N=85) | LJN452 140 μg (N=50) | LJN452 200 μg (N=51) | Placebo (N=97) | Total (N=350)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 5 | 2 | 4 | 15
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 3 | 8 | 14
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 6 | 2 | 3 | 15
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 3 | 3 | 5 | 15
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 4 | 3 | 7 | 6 | 22
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 2 | 2 | 8
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 2 | 3 | 4 | 13
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 5 | 2 | 2 | 10
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2 | 2 | 1 | 7
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 4 | 6 | 10 | 11 | 32
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 3 | 3 | 4 | 2 | 14
Fatigue (General disorders) | 0 | 3 | 1 | 5 | 7 | 3 | 9 | 28
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 6
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 3 | 0 | 6 | 10
Influenza (Infections and infestations) | 0 | 0 | 0 | 9 | 1 | 3 | 4 | 17
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 6 | 6 | 5 | 10 | 29
Periodontitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 5
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 3 | 0 | 7 | 11
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 8 | 9 | 3 | 10 | 32
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 9 | 0 | 3 | 14
Viral sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 5
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 3 | 1 | 3 | 3 | 10
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 4 | 4 | 2 | 12
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 6
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 1 | 2 | 1 | 9
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 2 | 1 | 1 | 7
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2 | 3 | 2 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 3 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 1 | 2 | 7 | 14
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3
Headache (Nervous system disorders) | 1 | 1 | 1 | 4 | 3 | 3 | 6 | 19
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0 | 4 | 3 | 2 | 11
Loss of libido (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 6
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 1 | 3 | 0 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 3 | 0 | 0 | 0 | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 7 | 26 | 35 | 15 | 88
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 5 | 3 | 4 | 15
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 4

LIMITATIONS AND CAVEATS:
No outputs were planned; and are not available for determining the effects of tropifexor on primary endpoints in the subset of patients who had historical biopsy data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT02855164/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT02855164/SAP_001.pdf